CLINICAL TRIAL: NCT01599130
Title: The Efficacy of Peg-interferon α-2a in HBeAg (+) Chronic Hepatitis B Patients Who Have Been Treated by Entecavir for 48 Weeks But Without HBeAg Loss
Brief Title: Efficacy of Peg-interferon α-2a in Hepatitis B Patients Treated by Entecavir Without HBeAg Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gao zhiliang, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhangyufeng
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; sequential peg-interferon-2a to entecavir
MeSH Terms: conditions — Hepatitis B | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- entecavir (Active Comparator): patients continue to use entecavir
  Interventions: Drug: Entecavir
- peg-interferon (Experimental): patients switch to sequential peg-interferon α-2a
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Entecavir — entecavir 0.5mg per day
  Other Names: Baraclude
  Arms: entecavir
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a 180ug per week
  Other Names: Pagasys
  Arms: peg-interferon

SUMMARY:
For HBeAg (+) hepatitis B patients who have been treated by entecavir for 48 weeks but without HBeAg loss, switching to peg-interferon may increase the response rate. In the investigators study, patients were divided into two groups. In Group A, patients continued entecavir for another 72 weeks. In Group B, patients switched to peg-interferon-2a monotherapy for 48 weeks, then followed up 24 weeks.

DETAILED DESCRIPTION:
For HBeAg positive hepatitis B patients who have been treated by entecavir for 48 weeks but without HBeAg loss, switching to peg-interferon may increase the response rate. In our study, patients without HBeAg loss to 48 weeks entecavir treatment were divided into two groups. In Group A, patients continued entecavir for another 72 weeks. In Group B, patients switched to peg-interferon-2a monotherapy for 48 weeks, then followed up 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old
* HBsAg(+) and HBeAg(+) for over 6 months before entecavir treatment
* Treated by entacavir for 48 weeks with HBeAg seroconversion

Exclusion Criteria:

* Pregnant women
* Decompensated liver disease
* Combination infection of HCV, HAV, or HEV
* Combination infection of HIV
* Any contraindication of interferon α

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
HBeAg sericonversion rate | 72 weeks

SECONDARY OUTCOMES:
HBeAg loss rate | 72 weeks
HBeAg quantification dynamic change | 72 weeks
HBsAg loss rate | 72 weeks
HBsAg seroconversion rate | 72 weeks
HBsAg quantification dynamic change | 72 weeks
ALT normalization rate | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhiliang Gao, Principal Investigator — The Third Affliated Hospital of Sun Yat-sen University
Locations (1):
- The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China